CLINICAL TRIAL: NCT04242940
Title: Assessing Listening Effort at Different Signal-to-noise Ratios in Bone-anchored Users
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The sponsor decided to terminate the study prematurely given that patient enrollment was delayed by more than two years relative to what originally stated in the protocol.
Sponsor: Oticon Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BC103
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Results first posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-04

CONDITIONS: Bilateral Hearing Loss
Keywords: Bone anchored hearing systems; BAHS; Listening effort; Pupillometry; Ponto 4
MeSH Terms: conditions — Hearing Loss, Bilateral

STUDY DESIGN:
Masking Description: The participants are however blinded to the Ponto 4 setting (OpenSound Navigator ON/OFF in Ponto 4) activated for each list of sentences.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ponto 4 sound processor (Experimental): All patients will be fitted with a bone-anchored sound processor (Ponto 4), unilaterally or bilaterally.
  Interventions: Device: Fitting of Ponto 4

INTERVENTIONS:
Device: Fitting of Ponto 4 — Bone-anchored hearing systems (BAHS) use the body's natural ability to transfer sound through bone conduction. The sound processor picks up sound and converts it into vibrations that are transferred through the skull bone to the inner ear (cochlea). Thus, for patients with conductive or mixed hearing losses, patients with lasting hearing loss following a middle ear disease or malformations (such as microtia), the vibrations are bypassing the conductive problem in the ear canal or middle ear. The intervention in this study is audiologically fitting one/two bone-anchored sound processors (Ponto 4) to patients that are already implanted with abutments.

SUMMARY:
The purpose of this study is to assess listening effort during a speech-in-noise task in bone-anchored hearing systems (BAHS) users via pupillometry.

DETAILED DESCRIPTION:
Pupil dilation can be used as an objective indicator of listening effort during the execution of a task. The aim is to compare listening effort with different settings (OpenSound Navigator ON and OFF) of Ponto 4, the sound processor released by Oticon Medical AB in June 2019, in listening scenarios that differ in complexity. The study consists of three visits of about two hours each in duration, during which the patients will perform a speech-in-noise task where the listening task varies in difficulty (i.e., in terms of signal-to-noise ratio, SNR). Pupil dilation will be recorded during the listening task as an indicator of listening effort. The patients will also use Ponto 4, instead of their own Ponto device, during a field-trial period of three months in between visit 2 and 3. Subjective evaluations of Ponto 4 will be performed via three questionnaires, one regarding self-reported performance in everyday life, one regarding work-related fatigue, and one regarding overall sound processor preference (Ponto 4 vs. patient's own device). All these outcome measures are non-invasive measurements. This is a post market study and all products used are CE marked and used in clinical practice worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 18 years and maximum 70 years old.
* UK English mother tongue.
* Bilateral conductive or mixed hearing loss.
* Users fitted unilaterally or bilaterally on abutment.
* Users are currently fitted with either Ponto 3, Ponto Plus or Ponto Pro (devices with a fitting range up to 45 dB HL).
* Users with at least 6 months of daily experience with one Ponto sound processor.
* BC thresholds of the implanted ear(s) better (lower) than or equal to 40 dB HL (average of 0.5, 1, 2 and 3 kHz) based on BC in-situ measurement at the first visit.
* People currently employed/self-employed (since the Need for Recovery questionnaire refers to work-related fatigue).
* Speech recognition scores better (higher) than or equal to 50% at +4 dB SNR with OSN OFF (as assessed via the first training list at Visit 1). This is to avoid including patients that are already "giving up" at +4 dB SNR.
* Users entitled for a sound-processor upgrade (according to the investigator) will first be selected. If there are not enough users entitled for an upgrade, then patients fitted with Ponto between 7 and 12 months before visit 1 will be considered. If there are not enough users within 7-12 months, then patients fitted with Ponto between 13 and 18 months before visit 1 will be considered.

Exclusion Criteria:

* Single-sided deafness (SSD)
* Hearing aid or cochlear implant on the opposite ear.
* Test persons with current eye diseases and/or history of eye surgery on both eyes.
* If the patient takes medications that can impact the autonomic nervous system - and hence pupil dilation (e.g., drugs for Parkinson's disease, peptic ulcers, incontinence, motion sickness).
* If the investigator or physician assesses that the patient is not fit for trial participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-02-21 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2022-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Brassington, Principal Investigator — University Hospitals Birmingham, United Kingdom
Locations (1):
- Audiology Department, Nuffield House, University Hospitals Birmingham, Birmingham, West Midlands, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ponto 4 Sound Processor
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ponto 4 Sound Processor
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.9 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Ponto fitting side [Number; unit: participants] — Ponto sound processor on the right side, left side, or both (bilateral).
  participants
    Right Side | 3
    Left Side | 2
    Bilateral | 8
BC in situ [Mean (Standard Deviation); unit: decibels] — Bone Conduction in situ - Pure tone average across .5, 1,2, & 3 kHz Population: BC in situ measures were not able to be obtained in 2 devices on the right ear and 3 on the left.
  decibels
    Right Ear: number analyzed (Participants) | 12
    Right Ear | 20.83 (9.82)
    Left Ear: number analyzed (Participants) | 11
    Left Ear | 22.61 (10.61)
PTA BC [Mean (Standard Deviation); unit: decibels] — Bone Conduction - Pure Tone average across .5, 1, 2, & 3kHz
  decibels
    Right Ear | 27.23 (9.62)
    Left Ear | 26.52 (9.53)
PTA AC [Mean (Standard Deviation); unit: decibels] — Air Conduction - Pure Tone average across .5, 1, 2, & 3 kHz
  decibels
    Right Ear | 63.75 (12.53)
    Left Ear | 61.96 (12.25)

OUTCOME MEASURES:

1. Primary Outcome: Overall Pupil Dilation
Description: Overall pupil dilation for OSN ON and OSN OFF at +4 dB SNR
  a third-order polynomial function was fit to the pupil dilation data, with the OSN setting as a fixed factor, as well as the interaction of OSN with each of the polynomial time terms. The formula used is the following: Pupil Dilation = (Linear + Quadratic + Cubic) X OSN setting + (1 + Linear + Quadratic + Cubic| Subject); where the Linear, Quadratic, and Cubic are the orthogonal terms; X indicates the interaction with OSN setting, and the terms reported in the second parenthesis are the random factors. The random factors include the effect of listeners, and of each of the time terms, to account for the variability in the time course of dilation across listeners.
  Outcome measure is the percentage reduction(% change) in pupil dilation with OSN ON vs OSN OFF
Time Frame: 10 days
Population: Four subjects had too many eye blinks in their pupillometry recordings (>15% of trials) and therefore their pupil data were unable to be analyzed.
  Note, ""OSN ON", "OSN OFF" are not two separate arms/groups. "OSN ON", "OSN OFF" are test conditions.
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | Ponto 4 Sound Processor
Number analyzed (Participants) | 10
percentage change | 58.7 (0.3)

2. Secondary Outcome: Peak Pupil Dilation (PPD) for OSN ON and OSN OFF
Description: The difference in pupil dilation between OSN ON and OSN OFF was also analyzed via Peak Pupil Dilation (PPD); thus, by investigating differences in dilation at the peak of the curve. The PPD was obtained for each subject as the maximum dilation between 7.5 and 9 s.
Time Frame: 10 days
Population: Four subjects had too many eye blinks in their pupillometry recordings (>15% of trials) and therefore their pupil data were unable to be analyzed.
Measure: Mean (Standard Deviation); unit: Arbitrary units
Arm/Group | Ponto 4 Sound Processor
Number analyzed (Participants) | 10
Arbitrary units
  PPD - OSN OFF | 1.80 (1.34)
  PPD - OSN ON | 1.05 (1.56)

3. Secondary Outcome: Speech Recognition Scores With OSN ON vs. OSN OFF Across SNRs
Description: A mixed-linear model with OSN setting (2 levels: ON and OFF) and SNR (5 levels: -8, -4, 0, +4, +8 dB) as fixed factors, and subject as random factor, was fit to the data.
Time Frame: 10 days
Population: Note that one subject did not perform the measurement at 0 dB SNR for OSN ON. Hence, the mean and std for OSN ON at 0 dB SNR is calculated for N=13, while all the other conditions are averaged across all subjects (N=14).
Measure: Mean (Standard Deviation); unit: Percentage correct
Arm/Group | Ponto 4 Sound Processor
Number analyzed (Participants) | 14
Percentage correct
  OSN ON -8dB SNR | 21.66 (16.24)
  OSN ON -4dB SNR | 51.77 (19.63)
  OSN ON 0dB SNR: number analyzed (Participants) | 13
  OSN ON 0dB SNR | 79.26 (13.96)
  OSN ON +4dB SNR | 95.41 (3.33)
  OSN ON +8dB SNR | 97.41 (2.49)
  OSN OFF -8dB SNR | 5.82 (8.27)
  OSN OFF -4dB SNR | 30.85 (25.61)
  OSN OFF 0dB SNR | 66.51 (16.31)
  OSN OFF +4dB SNR | 89.45 (6.38)
  OSN OFF +8dB SNR | 95.78 (3.95)

4. Secondary Outcome: Speech Spatial and Qualities of Hearing Scale (SSQ) Questionnaire Scores
Description: Self-reported perception before, during (at 1 month), and after field trial (at 3months).
  The SSQ questionnaire consists of 49 items with a scale from 0-10 where 0 represents "Not at all" and 10 represents "Perfect".
  The SSQ questionnaire is comprised of three subscales domains (Speech, Spatial, and Qualities of Hearing) - that is, each of the 49 items fits into one of these subscale "categories".
  The subscale scores AND the total scores (the total score is comprised of all of the 49 items) use the same scale of 0 to 10 where 0 represents "Not at all" and 10 represents "Perfect". For the total scale and all subscales (again all questions and by extension, the scales range from 0 to 10) the higher the value (closer to 10) represents a better outcome than lower values (closer to 0).
Time Frame: 4 months
Population: Two subjects did not complete the SSQ at the 1 month timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ponto 4 Sound Processor
Number analyzed (Participants) | 14
score on a scale
  Before Trial - Speech | 4.98 (1.60)
  Before Trial - Spatial | 3.87 (1.35)
  Before Trial - Qualities | 5.98 (1.63)
  Before Trial - Total | 4.94 (1.33)
  1 month - Speech: number analyzed (Participants) | 12
  1 month - Speech | 5.67 (1.46)
  1 month - Spatial: number analyzed (Participants) | 12
  1 month - Spatial | 4.87 (1.66)
  1 month - Qualities: number analyzed (Participants) | 12
  1 month - Qualities | 6.67 (1.13)
  1 month - Total: number analyzed (Participants) | 12
  1 month - Total | 5.74 (1.34)
  3 months - Speech | 5.88 (1.35)
  3 months - Spatial | 4.83 (1.45)
  3 months - Qualities | 6.46 (1.12)
  3 months - Total | 5.72 (1.23)

5. Secondary Outcome: Preference Questionnaire Scores.
Description: Self-reported preference after field trial. The preference questionnaire consists of 11 questions. The scores are from 1 to 5, where 1 means "Own sound processor much better" and 5 means "Test sound processor [Ponto 4] much better".
Time Frame: 4 months
Population: One subject did not complete the preference questionnaire.
Measure: Number; unit: participants
Arm/Group | Ponto 4 Sound Processor
Number analyzed (Participants) | 13
participants
  Prefer Ponto 4 | 11
  No preference | 2
  Prefer own device | 0

6. Secondary Outcome: Aided Sound Field Thresholds
Description: Sound field audiometry performed with the Auricle system while the patient is wearing the Ponto sound processor. This measurement is conducted at 10 frequencies from 250 Hz to 8 kHz. The Pure tone threshold is calculated as the average across .5, 1, 2, & 3 kHz)
Time Frame: 4 months
Population: A threshold was unable to be obtained for two subjects' right ears and three left ears.
Measure: Mean (Standard Deviation); unit: decibels
Arm/Group | Ponto 4 Sound Processor
Number analyzed (Participants) | 14
decibels
  Aided Right Ear: number analyzed (Participants) | 12
  Aided Right Ear | 32.29 (9.35)
  Aided Left Ear: number analyzed (Participants) | 11
  Aided Left Ear | 37.95 (9.12)

7. Secondary Outcome: BC in Situ Thresholds.
Description: Hearing level thresholds (dB HL) as assessed in situ with Ponto 4 placed on the patient's abutment. Bone-conduction thresholds (BC) are measured as the softest sound level that is audible by the patient at 10 frequencies from 250 Hz to 8 kHz. The Pure tone threshold is calculated as the average across .5, 1, 2, & 3 kHz
Time Frame: 1 hour
Population: A threshold was unable to be obtained for two subjects' right ears and three left.
Measure: Mean (Standard Deviation); unit: decibels
Arm/Group | Ponto 4 Sound Processor
Number analyzed (Participants) | 14
decibels
  BC in situ Right Ear: number analyzed (Participants) | 12
  BC in situ Right Ear | 20.83 (9.82)
  BC in situ Left Ear: number analyzed (Participants) | 11
  BC in situ Left Ear | 22.61 (10.61)

8. Other Pre Specified Outcome: Need for Recovery (NFR) Questionnaire Scores.
Description: Self-reported work-related fatigue. The NFR scale is an 11-item scale assessing the effects of fatigue caused by work (e.g., " I find it hard to relax at the end of a working day"). Possible responses are "yes" or "no". The total NFR score is the number of "yes" responses divided by the total number of items, presented as a percentage (i.e., range 0-100). The higher the score, the greater the NfR felt by the respondent. Scores with own device compared with Ponto 4 after 3months field trial are reported.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ponto 4 Sound Processor
Number analyzed (Participants) | 14
score on a scale
  Own device | 47.4 (37.3)
  Ponto 4 (3 months) | 47.4 (34.0)

9. Other Pre Specified Outcome: Pupil Dilation After Field Trial.
Description: Change in pupil dilation after field trial to check for acclimatization effects. Comparison of speech recognition scores for OSN Auto and OSN OFF at start and end of field trial.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: percent correct speech scores
Arm/Group | Ponto 4 Sound Processor
Number analyzed (Participants) | 14
percent correct speech scores
  OSN Auto at start | 94.7 (5.1)
  OSN Auto at end | 94.4 (2.7)
  OSN OFF at start | 89.5 (6.4)
  OSN OFF at end | 86.9 (7.6)

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Ponto 4 Sound Processor
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

LIMITATIONS AND CAVEATS:
Oticon Medical decided to terminate the study prematurely leading to a small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-11): https://cdn.clinicaltrials.gov/large-docs/40/NCT04242940/Prot_SAP_000.pdf